CLINICAL TRIAL: NCT04258943
Title: A Phase I/II Study of Bosutinib in Pediatric Patients With Newly Diagnosed Chronic Phase or Resistant/Intolerant Ph + Chronic Myeloid Leukemia", Study ITCC-054/COG-AAML1921
Brief Title: Bosutinib in Pediatric Patients With Newly Diagnosed Chronic Phase or Resistant/Intolerant Ph + Chronic Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: Erasmus Medical Center (Other); Dutch Childhood Oncology Group (Other); Innovative Therapies for Children with Cancer (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML1921; ITCC-054 (Registry Identifier: ITCC); 2015-002916-34 (EudraCT Number); 2023-504311-32-00 (Other: EU CT Number); NTR5501 (Other: NTR)
Record Dates: First submitted 2020-01-16; First posted 2020-02-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Philadelphia Chromosome Positive CML; Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Chronic Phase Chronic Myelogenous Leukemia
Keywords: Philadelphia Chromosome Positive CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Agent Bosutinib (Experimental): Bosutinib administered orally once daily in pediatric patients with newly diagnosed chronic phase Ph+ CML (ND CML) and pediatric patients with Ph+CML who have received at least one prior TKI therapy (R/I CML). A treatment cycle is defined as 28 days
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Patients with R/I disease are enrolled at a dose of 400 mg/m2 (DL2B) based on tolerability and PK analysis. Once the RP2D for R/I patients (RP2DR/I) is determined in the Phase 1, subsequent patients with R/I disease will be enrolled at the RP2DR/I for this subpopulation for the Phase 2 component of the study (see section 1.6.3 and section 3 for details).
  - Patients with newly diagnosed disease are being enrolled on Phase 2 component only, at RP2DND dose of 300 mg/m2. (see section 1.6.3 and section 3 for details)

SUMMARY:
This is a Phase 1-2, multicenter, international, single-arm, open-label study designed to identify a recommended dose of bosutinib administered orally once daily in pediatric patients with newly diagnosed chronic phase Ph+ CML (ND CML) and pediatric patients with Ph+CML who have received at least one prior TKI therapy (R/I CML), to preliminary estimate the safety and tolerability and efficacy, and to evaluate the PK of bosutinib in this patient population.

DETAILED DESCRIPTION:
The Phase 1 part of the study employs a 6+4 design (no DLT in 6 patients or 1 DLT in 10 patients) and incorporates additional PK information before escalating to the next dose level. If there is unacceptable toxicity or if PK results have exceeded the acceptable exposure levels for the adult equivalent dose, further dose escalation will be prohibited. The Recommended Phase 2 Dose (RP2D) is defined as the dose that results in equivalent(approximately ±20% of the adult values) PK exposure to 500 mg/day in adults and with 0 of 6 or <2 DLTs observed out of 10 evaluable patients with Ph+ CML and resistance or intolerance to prior TKI therapy. The phase 2 part of the study will enroll the following patient populations.

* Newly diagnosed (ND): newly diagnosed pediatric Ph + CML patients in chronic phase (CP)
* Resistant/intolerant (R/I): chronic phase or advanced (accelerated (AP) or blast phase (BP) pediatric Ph+ CML patients with resistance or intolerance to at least 1 prior TKI

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria Phase 1 (R/I patients only)

1. Cytogenetic and molecular diagnosis of Philadelphia chromosome-positive CML[2] at either time of initial CML diagnosis or at time of study screening:

   Cytogenetics must be performed by chromosome banding analysis (CBA) of bone marrow cell metaphases, and requires at least 20 metaphases.

   Only if dividing marrow cells cannot be obtained, or if there is an insufficient number of metaphases, CBA can be substituted by interphase fluorescence in situ hybridization (I-FISH) of bone marrow or peripheral blood cells, using dual color dual fusion probes, that allow the detection of BCR-ABL+ nuclei; at least 200 nuclei should be counted.

   Qualitative RT-PCR should be performed on RNA extracted from freshly collected bone marrow or peripheral blood cells. It identifies the transcript type, either e14a2 or 13a2 (also known as b3a2 and b2a2), or much more rarely e19a2, or e1a2, indicating the BCRABL protein weight (P210, rarely P230 or P190).
2. Resistance (suboptimal response or failure, as defined by 2013 European Leukemia Net guidelines[3]) or intolerance (with or without suboptimal response or failure) to at least one prior tyrosine kinase inhibitor (TKI) The 2013 European LeukemiaNet guidelines[3] will be used to define suboptimal response and failure to prior TKI therapy. Details are provided in appendices 3 (intolerance or failure after one TKI) and 4 (Failure after more than one TKIs).

   Intolerance to prior TKI therapy will be determined by the treating investigator, but generally applies to patients who are unable to receive standard or reduced doses of a TKI due to significant drug-related toxicity and/or when the drug-related toxicity is not responding to appropriate medical management. Patients who enroll as a result of intolerance to prior TKI therapy may have any level of response to their prior therapy and still be eligible.
3. Age ≥1 and <18 years at day of attaining the informed consent.
4. Lansky performance status ≥50% for patients ≤16 years of age, or Karnofsky scale ≥50% for patients >16 years of age (appendix 5).
5. Adequate bone marrow function:

   For second-line and third-line CP CML patients:

   Absolute neutrophil count >1000/mm3 (>1.0 x109/L); Platelets ≥75,000/mm3 (≥75 x109/L) without any platelet transfusions during the preceding 7 days.

   For fourth-line CP and all for all AP/BP CML patients:

   Absolute neutrophil count >500/mm3 (>0.5 x109/L); Platelets ≥50,000/mm3 (≥50 x109/L) without any platelet transfusions during the preceding 7 days.
6. Adequate Renal Function: Subjects must have a calculated creatinine clearance (CrCl) ≥ 60mL/min/1.73 m2, using the Schwartz formula to estimate GFR (see appendix 11).
7. Adequate liver function, including:

   AST/ALT ≤2.5 x upper limit normal (ULN) or ≤5 x ULN if attributable to disease involvement of the liver; Total bilirubin ≤1.5 x ULN unless the patient has documented Gilbert syndrome.
8. Recovered to Grade 0-1, or to baseline, from any acute toxicities of prior chemotherapy, immunotherapy, radiotherapy, differentiation therapy, or biologic therapy, with the exception of alopecia.
9. Able to reliably swallow whole capsules, whole tablets; or drug added to a suitable foodstuff (from capsule contents, added to either apple sauce or yoghurt); or tablets and/or capsules dissolved in water as an oral syringe drinking solution, or tablets dissolved and administered by NG tube when needed.
10. Serum/urine pregnancy test (for all girls ≥ age of menarche) negative at screening.
11. Male and female patients of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active.
12. Written informed consent of parent(s)/legal guardian(s) and/or patients (when applicable depending on age and local law and regulations)
13. Patients (including legally acceptable representative for minors where applicable) who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion criteria Phase 1 (R/I patients only)

Patients presenting with any of the following will not be included in the study:

1. Diagnosis of primary Ph+ acute lymphoblastic leukemia.
2. In patients with AP/BP CML: leptomeningeal leukemia, defined as positive cytology on lumbar puncture (including both CNS2 and CNS3 status), or clinical symptoms or signs present. This assessment is not required for inclusion of CP CML patients.
3. Extramedullary disease only.
4. Documented prior history of T315I or V299L BCR-ABL1 mutations (Note: BCR-ABL1 mutation testing will be performed at screening for a baseline assessment, but results are not used to determine eligibility. This exclusion criterion is based on whether there is a known history of these mutations at the time of study entry. If these mutations become evident during the study the patient will go off study).
5. Any prior treatment with a TKI within 7 days prior to starting bosutinib treatment, or other antitumor or anti-leukemia treatment (with the exception of hydroxyurea and/or anagrelide) within 14 days prior to start of bosutinib treatment.
6. Prior growth factors or biologic agents within 7 days prior to bosutinib treatment.
7. Use of strong or moderate CYP3A4 inhibitors and inducers (see Appendix 8) within 7 days prior and/or concomitant to bosutinib treatment
8. Use of proton pump inhibitors (Ph-modifying agents) within 7 days prior and/or concomitant to bosutinib treatment.
9. Prior radiotherapy within 3 months prior to bosutinib treatment.
10. Allogeneic stem cell transplantation within 3 months prior to bosutinib treatment.
11. Donor lymphocyte infusion (DLI) within 1 month prior to bosutinib treatment.
12. Hereditary bone marrow failure disorder.
13. Graft-versus-host disease (GVHD) within 60 days prior to bosutinib treatment.
14. Major surgery within 14 days prior to bosutinib treatment (recovery from any previous surgery should be complete before day 1).
15. History of clinically significant or uncontrolled cardiac disease, including:

    History of or active congestive heart failure; Clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); Diagnosed or suspected congenital or acquired prolonged QT syndrome; History of prolonged QTc.
16. Prolonged QTc (>450 msec, average of triplicate ECGs).
17. Need for medications known to prolong the QT interval.
18. Pregnant and/or nursing women
19. Uncorrected hypomagnesemia or hypokalemia due to potential effects on the QT interval.
20. Left ventricular ejection fraction <50% or shortening fraction <28%.
21. Recent or ongoing clinically significant gastrointestinal disorder that may interfere with the intake or absorption of the drug.
22. Evidence of serious active or uncontrolled bacterial, fungal or viral infection.
23. Known history of hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
24. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Inclusion criteria Phase 2

* Resistant/Intolerant CML patients: R/I The inclusion criteria for the R/I patients in Phase 2 are identical to the Phase 1 inclusion criteria.
* Newly Diagnosed CML patients

  1. Cytogenetic and molecular diagnosis of Philadelphia chromosome-positive CML at either time of initial CML diagnosis or at time of study screening:

     Cytogenetics must be performed by chromosome banding analysis (CBA) of bone marrow cell metaphases, and requires at least 20 metaphases.

     Only if dividing marrow cells cannot be obtained, or if there is an insufficient number of metaphases, CBA can be substituted by interphase fluorescence in situ hybridization (I-FISH) of bone marrow or peripheral blood cells, using dual color dual fusion probes, that allow the detection of BCR-ABL+ nuclei; at least 200 nuclei should be counted.

     Qualitative RT-PCR should be performed on RNA extracted from freshly collected bone marrow or peripheral blood cells. It identifies the transcript type, either e14a2 or e13a2 (also known as b3a2 and b2a2), or much more rarely e19a2, or e1a2, indicating the BCRABL protein weight (P210, rarely P230 or P190).
  2. Newly diagnosed CP Ph+ CML of ≤ 6 months (from initial diagnosis) without any previous TKI treatment (with the exception of hydroxyurea and/or anagrelide) for CML. Diagnosis of CP CML will be defined as per Appendix 1.
  3. Age ≥1 and <18 years at day of attaining the informed consent.
  4. Lansky performance status ≥50% for patients ≤16 years of age, or Karnofsky scale ≥50% for patients >16 years of age (appendix 5).
  5. Adequate Renal Function: Subjects must have a calculated creatinine clearance (CrCl) ≥ 60 mL/min/1.73 m2, using the Schwartz formula to estimate GFR (see appendix 11).
  6. Adequate liver function, including:

     AST/ALT ≤2.5 x upper limit normal (ULN) or ≤5 x ULN if attributable to disease involvement of the liver; Total bilirubin ≤1.5 x ULN unless the patient has documented Gilbert syndrome.
  7. Able to reliably swallow whole capsules, whole tablets; or drug added to a suitable foodstuff (from capsule contents, added to either apple sauce or yogurt); or tablets and/or capsules dissolved as an oral syringe drinking solution, or tablets dissolved and administered by NG tube when needed.
  8. Serum/urine pregnancy test (for all girls ≥ age of menarche) negative at screening.
  9. Male and female patients of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active.
  10. Written informed consent of parent(s)/legal guardian(s) and/or patients (when applicable depending on age and local law and regulations)
  11. Patients (including legally acceptable representative for minors where applicable) who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion criteria Phase 2

* Resistant/Intolerant (R/I) CML patients: The exclusion criteria for the R/I cohort in Phase 2 are identical to the Phase 1 exclusion criteria.
* Newly Diagnosed CML patients:

Patients presenting with any of the following will not be included in the study:

1. Diagnosis of primary Ph+ acute lymphoblastic leukemia.
2. Extramedullary disease only.
3. Documented prior history of T315I or V299L BCR-ABL1 mutations (Note: BCR-ABL1 mutation testing will be performed at screening for a baseline assessment, but results are not used to determine eligibility. This exclusion criterion is based on whether there is a known history of these mutations at the time of study entry. If these mutations become evident during the study the patient will go off study).
4. Any prior treatment with a TKI or other anti-tumor or anti-leukemia treatment (with the exception of hydroxyurea and/or anagrelide)
5. Prior growth factors or biologic agents within 7 days prior to bosutinib treatment.
6. Use of strong or moderate CYP3A4 inhibitors and inducers (see Appendix 8) within 7 days prior and/or concomitant to bosutinib treatment
7. Use of proton pump inhibitors (Ph-modifying agents) within 7 days prior and/or concomitant to bosutinib treatment)
8. Hereditary bone marrow failure disorder.
9. Major surgery within 14 days prior to bosutinib treatment (recovery from any previous surgery should be complete before day 1).
10. History of clinically significant or uncontrolled cardiac disease, including:

    * History of or active congestive heart failure;
    * Clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
    * Diagnosed or suspected congenital or acquired prolonged QT syndrome;
    * History of prolonged QTc.
11. Prolonged QTc (>450 msec, average of triplicate ECGs).
12. Need for medications known to prolong the QT interval.
13. Pregnant and/or nursing women
14. Uncorrected hypomagnesemia or hypokalemia due to potential effects on the QT interval.
15. Left ventricular ejection fraction <50% or shortening fraction <28%.
16. Recent or ongoing clinically significant gastrointestinal disorder that may interfere with the intake or absorption of the drug.
17. Evidence of serious active or uncontrolled bacterial, fungal or viral infection.
18. Known history of hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
1. Incidence (and severity) of Dose-Limiting Toxicities (DLTs) assessed during the first 28 days of treatment. | First 28 days of treatment (first cycle)
  Data from Phase 1; Dose-limiting toxicities determined as adverse events occurring in the first cycle (28 days) of treatment, which are attributable to bosutinib. Assessment will be done according the following DLT definition:
  * Non-hematologic AEs: grade ≥3 toxicities, except those that have not been optimally treated; any grade ≥2 toxicity requiring discontinuation/interruption for ≥7 days during the first 28 days of treatment; clinically significant laboratory abnormalities grade ≥3 or lasting ≥7 days despite optimal treatment
  * Hematologic AEs: grade 4 neutropenia or thrombocytopenia lasting ≥7 days (not explained by persistent leukemia).
PK parameters of bosutinib: Maximum observed plasma concentration (Cmax) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose and before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days); unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 1; Maximum plasma concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time postdose and actual dose will be used for all calculations.
PK parameters of bosutinib:Time to Cmax (Tmax) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 1; Time to maximum plasma concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post dose and actual dose will be used for all calculations.
PK parameters of bosutinib: Area under the plasma concentration versus time curve from time zero to the dosing interval (AUCτ) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 1; Area under the plasma concentration versus time curve from time zero to the dosing interval calculated from the plasma concentration-time data by linear trapezoidal rule during the ascending phase and log trapezoidal rule during the descending phase.
PK parameters of bosutinib: Pre-dose concentration (Ctrough) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 1; Pre-dose concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post dose and actual dose will be used for all calculations.
PK parameters of bosutinib: Apparent clearance (CL/F). | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 1; Apparent clearance of the drug from plasma after oral administration, calculated as Dose/AUCt.
AEs, as characterized by type, frequency, severity (as graded using CTCAE version, v4.03), timing, seriousness, and relation to study therapy (pooled across ND and R/I CML patients and by line of therapy). | AE's will be collected from signing informed consent continuously during the study until 28 days after last dose (on average, 2 years).
  Data from Phase 2; AEs will be graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA). Treatment emergent AEs (TEAEs) are defined as those with initial onset or increasing in severity after the first dose of study medication. Endpoints include maximum toxicity, time to first event (time from first dose to date of first event including only non-partial dates), duration of any stage/grade event (time from start date to stop date including only non-partial dates).
PK parameters of bosutinib: Maximum observed plasma concentration (Cmax) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose and before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 & and before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 2; subset of newly diagnosed patients. Maximum plasma concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post-dose and actual dose will be used for all calculations.
PK parameters of bosutinib:Time to Cmax (Tmax) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 2; subset of newly diagnosed patients. Time to maximum plasma concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post-dose and actual dose will be used for all calculations.]
PK parameters of bosutinib: Area under the plasma concentration versus time curve from time zero to the dosing interval (AUCτ) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 2; subset of newly diagnosed patients. Area under the plasma concentration versus time curve from time zero to the dosing interval calculated from the plasma concentration-time data by linear trapezoidal rule during the ascending phase and log trapezoidal rule during the descending phase.
PK parameters of bosutinib: Pre-dose concentration (Ctrough) | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 2; subset of newly diagnosed patients. Pre-dose concentration of bosutinib calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post-dose and actual dose will be used for all calculations.
PK parameters of bosutinib: Apparent clearance (CL/F). | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing (each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase 2; subset of newly diagnosed patients. Apparent clearance of the drug from plasma after oral administration, calculated as Dose/AUCt.
Population PK parameters of bosutinib including volume of distribution based on combined PK data from Phase 1 and Phase 2 | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose & before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing(each cycle is 28 days); for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase1 and Phase 2. Population PK parameters of bosutinib including volume of distribution based on combined PK data from Phase 1 and Data from Phase1 and Phase 2. Volume of distribution are calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post-dose and actual dose will be used for all calculations.
Population PK parameters of bosutinib including clearance based on combined PK data from Phase 1 and Phase 2 | Cycle 1 Day 14: pre-dose & 1, 3, 6, 8, & 24 hours post-dose and before day 15 dosing; Cycles 2, 3 & 4, Day 1: 24 hours post Day 14 dose & before Day 15 dosing(each cycle is 28 days);for unexpected and/or serious bosutinib-related AEs: when AE is detected
  Data from Phase1 and Phase 2. Clearance is calculated from the plasma concentration-time data using noncompartmental analysis (NCA). The calculated elapsed time post-dose and actual dose will be used for all calculations

SECONDARY OUTCOMES:
AEs, as characterized by type, frequency, severity (as graded using CTCAE version, v4.03), timing, seriousness, and relation to study therapy; | From signing informed consent, continuously during the study until 28 days after last dose (on average 2 years).
  Data from Phase 1. AEs will be graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA). Treatment emergent AEs (TEAEs) are defined as those with initial onset or increasing in severity after the first dose of study medication. Endpoints include maximum toxicity, time to first event (time from first dose to date of first event including only non-partial dates), duration of any stage/grade event (time from start date to stop date including only non-partial dates).]
Occurrence of laboratory abnormalities of hematology, blood chemistry, liver functions, coagulation, HbsAg, urinalysis and pregnancy tests values, as characterized by type, frequency, severity and timing summarized in an overview table | Screening; cycle 1 days 1, 8, 14, 22; cycles 2 to 7: at start of every cycle; cycle 8 and higher: every 3 cycles; End of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 1. Test abnormalities in hematology, blood chemistry, liver functions, coagulation, HbsAg, urinalysis and pregnancy test will be recorded. Severity of laboratory test abnormalities will be graded using NCI CTCAE version, v4.03. For those laboratory abnormalities without CTCAE grade definitions, results will be categorized as normal, abnormal or not done. Coagulation and HBsAG only tested at screening. Urinalysis and pregnancy test and contraception check not tested at days 8, 14, 15 and 22 of cycle 1. Urinalysis not performed at beginning of cycles 2, 3, 5 and 6
ECG abnormalities: QT interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 1. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points. Kamofsky or Lansky performance score is collected to evaluate performance status.
ECG abnormalities: RR interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 1. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points.
ECG abnormalities: PR interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 1. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points.
ECG abnormalities: QRS duration | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 1. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points.
Performance status abnormalities | Screening; on day 1 of every subsequent cycle end of treatment (each cycle is 28 days)
  Data from Phase 1. Kamofsky or Lansky (depending on age) performance score as assessed by physician is collected to evaluate performance status
Overall cumulative disease response: complete hematologic response (CHR), major cytogenetic response (MCyR), major molecular response (MMR) and deep molecular response | Hematologic response:Screening; Cycles 2 to 7: start of every cycle; cycle 8 and higher: every 3 cycles; End of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1. MCyR is defined as complete cytogenetic response [CCyR] plus partial cytogenetic response [PCyR]. (definitions in appendix 2).]
Overall cumulative disease response: complete hematologic response (CHR), major cytogenetic response (MCyR), major molecular response (MMR) and deep molecular response | Screening; Cycles 2 to 7: start of every cycle; cycle 8 and higher: every 3 cycles; End of treatment: within 28 days after last dose (each cycle is 28 days).]
  Data from Phase 2. MCyR is defined as complete cytogenetic response [CCyR] plus partial cytogenetic response [PCyR]. (definitions in appendix 2).
Time to the respective responses by line of therapy | Through study completion, a maximum of around 10 years
  Time to response is defined as the time period from start of treatment with bosutinib to first response, unconfirmed for molecular and cytogenetic and confirmed for hematologic. Patients without events are censored at the last molecular, cytogenetic, or hematologic assessment where response could be assessed for the respective endpoint
Duration of the respective responses by line of therapy | Through study completion, a maximum of around 10 years
  Data from Phase 2. Duration of response is defined is defined as the time period from the date of the earliest demonstration of a response until the earliest date of confirmed loss of that response.
Event-free survival (EFS; including time to transformation to AP and BP CML) by line of therapy (definition in appendix 2). | Through study completion, a maximum of around 10 years
  Data from Phase 2. EFS is defined as the interval from the date of first dose of bosutinib until the earlier date of EFS events. Patients without the event will be censored at the last evaluation date.
Overall survival (OS) in pediatric patients with Ph+ CML by line of therapy | Through study completion, a maximum of around 10 years
  Data from Phase 2. OS or survival time is defined as the interval from the date of first dose of bosutinib until the date of death due to any cause. Patients without the event will be censored at the last evaluation date
Occurrence of laboratory abnormalities of hematology, blood chemistry, liver functions, coagulation, HbsAg, urinalysis and pregnancy tests values, as characterized by type, frequency, severity and timing summarized in an overview table | Screening; cycle 1 days 1, 8, 14, 22; cycles 2 to 7: at start of every cycle; cycle 8 and higher: every 3 cycles; End of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 2. Pooled across ND and R/I CML and by line of therapy. Test abnormalities in hematology, blood chemistry, liver functions, coagulation, HbsAg, urinalysis and pregnancy test and contraception will be recorded. Severity of laboratory test abnormalities will be graded using NCI CTCAE version, v4.03. For those laboratory abnormalities without CTCAE grade definitions, results will be categorized as normal, abnormal or not done. Coagulation and HBsAG only tested at screening. Urinalysis and pregnancy test and contraception check not tested at days 8, 14, 15 and 22 of cycle 1. Urinalysis not performed at beginning of cycles 2, 3, 5 and 6
ECG abnormalities: QT interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 2. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points
ECG abnormalities: RR interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 2. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points
ECG abnormalities: PR interval | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 2. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points
ECG abnormalities: QRS duration | For ECG: Screening; Cycle 1, day 14; Cycles 2, 3 and 4, day 1; end of treatment: within 28 days after last dose (each cycle is 28 days)
  Data from Phase 2. ECG measurements (an average of the triplicate measurements) will be used for the statistical analysis and all data presentations. Any data obtained from ECGs repeated for safety reasons after the nominal time points will not be averaged along with the preceding triplicates. Interval measurements from repeated ECGs will be included in the outlier analysis (categorical analysis) as individual values obtained at unscheduled time points
Performance status abnormalities | Screening; on day 1 of every subsequent cycle end of treatment (each cycle is 28 days)
  Data from Phase 2. Kamofsky or Lansky (depending on age) performance score as assessed by physician is collected to evaluate performance status.

OTHER OUTCOMES:
Parameters of bone metabolism and growth: linear growth | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX). The analysis of bone age, pubertal status and results of serum chemistry tests will be descriptive. Height (cm), weight (kg), bone age (yr), Tanner stage, serum chemistry and bone densitometry scan results [Lumbar Spine (L1-L4) (g/cm2)] will be provided in listings and summarized by study visit (including change from baseline).
Parameters of bone metabolism and growth: bone age | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: bone mineral density of lumbar spine | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: physical signs of pubertal maturation (Tanner stage and testicular volume of boys), | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) | [Time Frame: Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: markers of bone formation and bone resorption (bone alkaline phosphatase and CTX). | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 1 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Patient and/or caregiver-reported assessments of gastrointestinal symptoms, as measured by selected domains from the Pediatric quality of life inventory ™ (PedsQL) Gastrointestinal Symptom Scale | Through study completion, a maximum of around 10 years
  Data from Phase 1. Pediatric quality of life inventory ™ (PedsQL) Gastrointestinal Symptom Scale questionnaires will be used to assess gastrointestinal symptoms. ON a scale of 0 to 4, with 0 being: 'never' and 4 being: 'almost always'
Patient and/or caregiver-reported assessment of the taste and ability to swallow the medicine, as measured by the Palatability Questionnaire for Bosutinib in patients aged 4-18 years of age. | Through study completion, a maximum of around 10 years
  Data from Phase 1. A questionnaire with different kind of questions, using a 1 to 3 score on difficulty to swallow, with 1 being' difficult to swallow' and 3 being:' no trouble, easy to swallow' and a 1 to 5 score on assessment of taste and overall ease, with 1 being: 'dislike very much' and 5 being: ' like very much'.
Parameters of bone metabolism and growth: linear growth | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX). The analysis of bone age, pubertal status and results of serum chemistry tests will be descriptive. Height (cm), weight (kg), bone age (yr), Tanner stage, serum chemistry and bone densitometry scan results [Lumbar Spine (L1-L4) (g/cm2)] will be provided in listings and summarized by study visit (including change from baseline).
Parameters of bone metabolism and growth: bone age | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: bone mineral density of lumbar spine | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: physical signs of pubertal maturation (Tanner stage and testicular volume of boys | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Parameters of bone metabolism and growth: markers of bone formation and bone resorption (bone alkaline phosphatase and CTX). | Screening; Start cycle 7; Cycle 8 and higher: every 12 months since start of therapy or every 6 months from cycle 7; end of treatment: within 28 days after last dose (each cycle is 28 days).
  Data from Phase 2 that includes linear growth, bone age, bone mineral density of lumbar spine, physical signs of pubertal maturation (Tanner stage and testicular volume of boys), and hormones associated with growth and pubertal development (IGF-1, T4, TSH and LH, FSH, estradiol for girls, and testosterone for boys) and a marker of bone formation and bone resorption (bone alkaline phosphatase and CTX).
Patient and/or caregiver-reported assessments of gastrointestinal symptoms, as measured by selected domains from the Pediatric quality of life inventory ™ (PedsQL) Gastrointestinal Symptom Scale. | Through study completion, a maximum of around 10 years
  Data from Phase 2. Pediatric quality of life inventory ™ (PedsQL) Gastrointestinal Symptom Scale questionnaires will be used to assess gastrointestinal symptoms. On a scale of 0 to 4, with 0 being: 'never' and 4 being: 'almost always'
Patient and/or caregiver-reported assessment of the taste and ability to swallow the medicine, as measured by the Palatability Questionnaire for Bosutinib in patients aged 4-18 years of age. | Through study completion, a maximum of around 10 years
  Data from Phase 2 A questionnaire with different kind of questions, using a 1 to 3 score on difficulty to swallow, with 1 being' difficult to swallow' and 3 being:' no trouble, easy to swallow' and a 1 to 5 score on assessment of taste and overall ease, with 1 being: 'dislike very much' and 5 being: ' like very much'.

CONTACTS AND LOCATIONS:
Locations (59):
- United States (45):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanene-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Specialty Center of Nevada II, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Lehigh Valley Hospital-Cedar Crest, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - CHU Lyon/Hospices Civils de Lyon, Lyon
  - Hopital Armand Trousseau, Paris
  - Hopital Robert Debré, Paris
- Universitätsklinikum Erlangen, Erlangen, Germany
- Italy (3):
  - San Gerardo Hospital, Monza
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Ospedale Regina Margerita, Torino
- Netherlands (2):
  - Erasmus Medical Center - Sophia Children's Hospital, Rotterdam
  - Prinses Maxima centrum voor kinderoncologie, Utrecht
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Niño Jesús, Madrid
- University Children's Hospital, Zurich, Switzerland
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - The Royal Marsden NHS Foundation Trust, London

REFERENCES:
- [Background] Baccarani M, Deininger MW, Rosti G, Hochhaus A, Soverini S, Apperley JF, Cervantes F, Clark RE, Cortes JE, Guilhot F, Hjorth-Hansen H, Hughes TP, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Martinelli G, Mayer J, Muller MC, Niederwieser D, Pane F, Radich JP, Rousselot P, Saglio G, Saussele S, Schiffer C, Silver R, Simonsson B, Steegmann JL, Goldman JM, Hehlmann R. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood. 2013 Aug 8;122(6):872-84. doi: 10.1182/blood-2013-05-501569. Epub 2013 Jun 26. PMID 23803709
- [Derived] Brivio E, Pennesi E, Willemse ME, Huitema ADR, Jiang Y, van Tinteren HDR, van der Velden VHJ, Beverloo BH, den Boer ML, Rammeloo LAJ, Hudson C, Heerema N, Kowalski K, Zhao H, Kuttschreuter L, Bautista Sirvent FJ, Bukowinski A, Rizzari C, Pollard J, Murillo-Sanjuan L, Kutny M, Zarnegar-Lumley S, Redell M, Cooper S, Bertrand Y, Petit A, Krystal J, Metzler M, Lancaster D, Bourquin JP, Motwani J, van der Sluis IM, Locatelli F, Roth ME, Hijiya N, Zwaan CM. Bosutinib in Resistant and Intolerant Pediatric Patients With Chronic Phase Chronic Myeloid Leukemia: Results From the Phase I Part of Study ITCC054/COG AAML1921. J Clin Oncol. 2024 Mar 1;42(7):821-831. doi: 10.1200/JCO.23.00897. Epub 2023 Nov 30. PMID 38033284
- See also: DutchTrial Register — https://onderzoekmetmensen.nl/en/trial/54687